CLINICAL TRIAL: NCT00682045
Title: A Prospective Observational Study of Usefulness of a T Cell-based Assay for Latent Tuberculosis Infection in Renal Transplant Recipients
Brief Title: Latent Tuberculosis Infection in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Sung-Han Kim, MD, Asan Medical Center
Other Study IDs: AMC-20080169
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-03

CONDITIONS: Renal Transplant
Keywords: tuberculosis; transplantation
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- T-SPOT.TB positive: T-SPOT.TB positive patients

SUMMARY:
The aim of this study is to estimate the usefulness of a T cell-based assay (i.e. T-SPOT.TB assay) for diagnosis of latent tuberculosis infection (LTBI) in renal transplant recipients. For this purpose, the investigators enrolled renal transplant recipients and observed the developement of tuberculosis within 1 to 2 years after the transplantation.

DETAILED DESCRIPTION:
We evaluate the usefulness of a newly-developed T cell-based assay prior to undergoing immunosuppression in renal transplant recipients. Among all renal transplant recipients, patients with negative tuberculin skin test and no other indications for latent tuberculosis infection will be enrolled in this study. We will exam T-SPOT.TB test in these patients, and observe the developement of tuberculosis within 1 to 2 years after the transplantation. The results of T-SPOT.TB will be blinded to the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or more
* Negative tuberculin skin test (induration less than 10 mm)

Exclusion Criteria:

* Recent contact of patients with active pulmonary tuberculosis
* Suspected active tuberculosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
development of tuberculosis | within 2 years after transplantation

SECONDARY OUTCOMES:
all cause mortality | within 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim SH, Lee SO, Park JB, Park IA, Park SJ, Yun SC, Jung JH, Kim YH, Kim SC, Choi SH, Jeong JY, Kim YS, Woo JH, Park SK, Park JS, Han DJ. A prospective longitudinal study evaluating the usefulness of a T-cell-based assay for latent tuberculosis infection in kidney transplant recipients. Am J Transplant. 2011 Sep;11(9):1927-35. doi: 10.1111/j.1600-6143.2011.03625.x. Epub 2011 Jul 12. PMID 21749641
- [Derived] Kim SH, Lee SO, Park IA, Park SJ, Choi SH, Kim YS, Woo JH, Park SK, Park JS, Kim SC, Han DJ. Diagnostic usefulness of a T cell-based assay for latent tuberculosis infection in kidney transplant candidates before transplantation. Transpl Infect Dis. 2010 Apr;12(2):113-9. doi: 10.1111/j.1399-3062.2010.00495.x. Epub 2010 Jan 25. PMID 20113458